CLINICAL TRIAL: NCT00285753
Title: Development and Evaluation of Support Groups for Patients With Mild Cognitive Impairment and Their Partners
Brief Title: Support Groups for Patients With Mild Cognitive Impairment and Their Partners
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Netherlands Alzheimer Foundation (Other)
Responsible Party: Department of medical psychology, UMCN St. radboud
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: V-2002-018; CMO-nr: 2003/071
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Mild Cognitive Impairment
Keywords: psychosocial intervention; mild cognitive impairment; support group; caregivers; Mild Cognitive Impairment (MCI); Cognitive Impairment No Dementia (CIND)
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: support groups — cognitive behavioral intervention with psychoeducation

SUMMARY:
This study aims at developing and evaluating a support group program for patients with mild cognitive impairment (MCI) and their partners. These patients have defective memory function but are not demented. However, there is an increased chance of developing dementia in the near future; 10-15% per year for MCI patients, in contrast to 1-2% per year for healthy elderly persons. For the patients and their caregivers this means that they are confronted with feelings of uncertainty and fear towards the future. They also have many questions about how to improve their memory problems and how to cope with other changes or consequences.

The purpose of the support group program is to improve coping skills and facilitate adaptation to the impairments, in order to reduce anxiety or depression and strengthen feelings of competence in patients and their partners.

DETAILED DESCRIPTION:
One of the consequences of the improved methodology for diagnosing dementia in a very early stage is a growing group of patients in memory clinics who have cognitive deficits, which exceed normal physiological aging processes but do not fulfil the criteria for dementia. This category of patients with so-called 'Mild cognitive impairment' (MCI) is known to have an increased risk at developing Dementia. For these patients, who have intact insight and expressive skills, we expect that a psychosocial intervention may reduce feelings of helplessness and anxiety and improve quality of life.

The group intervention was developed with respect to the 'stress adaptation coping model' of Lazarus and the 'family support model' of Bengston and Kuypers.

Coming up with these models the aim is to teach participants to explore their attributions, feelings and behaviour in order to enhance their coping strategies. This will increase the feelings of competence and decrease feelings of helplessness.

In addition to these models we investigated the problems and themes as they are experienced by MCI patients and their partners, using systematic interviews. This information resulted in the following modules:

1. Understanding MCI and memory problems;
2. Exploring attributions and misconceptions;
3. Other changes;
4. Methods to improve memory performance;
5. Worrying and problem solving;
6. Losing activities and finding a new balance;
7. Tension and relaxation;
8. Managing conflicts;
9. Emotions.

These modules are worked through in 10 sessions, in 12 weeks. The group structure is as follows: patients and parents meet separately the first 60 minutes, and then reconvene together for the last half hour. This structure optimizes the sharing of each other's experiences and prevents stigmatizing.

The main objective of the current study is to develop and evaluate a support group intervention for patients with MCI and their partners. We expect that our support group intervention will strengthen the partner's sense of competence to care for the patient and will improve the quality of life of the patient and the partner as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MCI (MCI criteria, Petersen, 2001 and Grundman, 2004) and their primary caregivers.

Exclusion Criteria:

* Mini-Mental State Examination (MMSE) < 23
* Severe mood disorder.
* No motivation.
* Severe language problems.
* Premorbid relationship problems

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2003-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
quality of life: RAND, GDS | pre and post treatment
caregiver: sense of competence (SCQ), burden of the problems in the Revised Memory and Behavioral Problems (RMBP) | pre- and post intervention

SECONDARY OUTCOMES:
Illness cognitions: Illness Cognitions Questionnaire (ICQ) | pre and post treatment
marital satisfaction: Maudsley Marital Questionnaire (MMQ) | pre and post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jan Pieter Teunisse, PhD, Principal Investigator — Radboud University Medical Center; Floor Kraaimaat, Professor, Principal Investigator — Radboud University Medical Center; Marcel Olde Rikkert, Professor, Principal Investigator — Coordinator Alzheimer Centre UMC Nijmegen; Myrra Vernooy, PhD, Principal Investigator — Coordinator Alzheimer Centre UMC Nijmegen
Locations (2):
- Netherlands (2):
  - Rijnstate Ziekenhuis, Arnhem, Gelderland
  - UMC Sint Radboud, Nijmegen, Gelderland

REFERENCES:
- [Derived] Banningh LW, Vernooij-Dassen MJ, Vullings M, Prins JB, Rikkert MG, Kessels RP. Learning to live with a loved one with mild cognitive impairment: effectiveness of a waiting list controlled trial of a group intervention on significant others' sense of competence and well-being. Am J Alzheimers Dis Other Demen. 2013 May;28(3):228-38. doi: 10.1177/1533317513481093. Epub 2013 Mar 25. PMID 23528880
- [Derived] Joosten-Weyn Banningh LW, Prins JB, Vernooij-Dassen MJ, Wijnen HH, Olde Rikkert MG, Kessels RP. Group therapy for patients with mild cognitive impairment and their significant others: results of a waiting-list controlled trial. Gerontology. 2011;57(5):444-54. doi: 10.1159/000315933. Epub 2010 Jul 20. PMID 20664181